CLINICAL TRIAL: NCT01875848
Title: Buprenorphine vs. Opioid Dose Escalation Among Patients With Chronic Pain
Acronym: Bup
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Data safety monitoring board recommended due to low recruitment yield.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPO 13-184
Record Dates: First submitted 2013-05-28; First posted 2013-06-12 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- buprenorphine/naloxone (Experimental): induction onto buprenorphine/naloxone from opioid treatment
  Interventions: Drug: buprenorphine/naloxone
- opioid dose escalation (Active Comparator): increase of up to 25% of current opioid dose
  Interventions: Drug: opioid dose escalation

INTERVENTIONS:
Drug: buprenorphine/naloxone — partial opioid agonist
  Other Names: Suboxone
  Arms: buprenorphine/naloxone
Drug: opioid dose escalation — up to 25% increase in patient's current opioid dose
  Other Names: No other names
  Arms: opioid dose escalation

SUMMARY:
This study compares buprenorphine/naloxone to opioid dose escalation among patients with poorly controlled non-cancer pain on 30-100 mg daily morphine equivalent opioid dose.

DETAILED DESCRIPTION:
Increasingly, Veterans are prescribed potent opioid analgesics for the treatment of chronic pain despite limited evidence for efficacy and increasing evidence of serious harms including addiction and non-fatal and fatal overdose. While guidelines recommend consideration of dose increase for patients not benefitting from opioid therapy, the rates of major harms are directly related to dose. Higher doses may also be more likely to precipitate opioid-induced hyperalgesia, a paradoxical increased pain response, in susceptible individuals. In summary, opioid dose increase, a currently accepted clinical response to poorly controlled pain, may offer little benefit and certainly increases risk, especially in patients already on moderate-high doses (30-100 mg daily morphine equivalents). Alternative treatment strategies to opioid dose escalation that lessen risk and possibly increase benefit are much needed.

Switching to buprenorphine/naloxone (BUP/NX), a partial opioid agonist approved for use in the treatment of opioid abuse/dependence, may be a safe and effective alternative strategy to opioid dose escalation in the treatment of chronic pain. As a partial agonist, there is a ceiling to BUP/NX's respiratory depressant and other opioid-like effects, meaning it is less likely to cause addiction and overdose. Additionally, there are pre-clinical data to suggest BUP/NX is less likely to produce opioid-induced hyperalgesia and may even reverse it in patients switched from full agonist opioids. Case series have demonstrated improvements in pain, functional status and quality of life among patients switched from full agonist opioids to BUP/NX for chronic pain. Controlled trials are needed to establish BUP/NX's efficacy compared to opioid dose escalation in the treatment of poorly-controlled pain.

The investigators propose a pilot 12-week, open label randomized trial of BUP/NX compared to opioid dose escalation among patients with poorly-controlled pain on the primary outcome of pain intensity. As patient acceptance of either opioid dose escalation or BUP/NX is unknown, the investigators' first objective is to assess willingness to enroll in a randomized trial and reasons for and against enrollment among eligible patients. The study will compare treatments on the primary outcome of pain intensity, measured using the 11-point pain numerical rating scale, and secondary outcomes of pain interference, using the Brief Pain Inventory functional interference subscale, medication adherence and patient global assessment of change. Mixed models will be employed in the analysis to accommodate potential unbalanced repeated measures with missing data. Effect size estimates will be used to generate sample size projections for a definitive trial. This line of research is a direct extension of the PI's HSR&D-funded CDA-2 project developing a screening tool to identify low efficacy opioid use in primary care and also well-aligned with the Strategic Plan and Focused Area of Research of the Pain Research, Informatics, Medical comorbidities, and Education (PRIME) Center's proposal for a Center of Innovation (COIN) and its strategic objective to "Promote access, continuity, and sustainability of safe and effective interventions for pain and pain-related disability."

ELIGIBILITY:
Participants were recruited and enrolled at VACT West Haven, CT. Participants are aged 18 and older and have 3 months or more of continuous opioid therapy for chronic pain. Participants are actively prescribed 30-100mg of morphine equivalent opioid dose based on pharmacy records. Primary Care Providers will assent for patient participation.

Inclusion Criteria:

* Aged 18 and older
* 3 months of continuous opioid therapy for chronic pain;
* 30-100 mg morphine equivalent daily opioid dose based on pharmacy records of standing and as needed opioids prescribed.
* 28 (out of 70) on the 7-item Brief Pain Inventory (BPI) functional interference subscale at screening
* Numerical pain rating of 4 or greater (i.e., moderate pain or greater) at screening on the 11-point pain numerical rating scale (NRS)
* Females must (a) be using birth control pills or depo provera injections, or have an intrauterine device; or (b) be post-menopausal, or (c) have undergone surgically sterilization.
* Primary care provider's (PCP) assent for patient participation, ascertained via encrypted email or in-person query.

Exclusion Criteria:

* DSM-IV defined substance use disorder, except nicotine dependence. Participants known to using marijuana, including those who are apparently legally authorized to use marijuana by non-VHA providers, will be excluded since opioid dose escalation in regular marijuana users is contraindicated.
* Opioid therapy for palliative care
* Participation in another investigational pharmaceutical trial within 30 days of screening
* Pregnancy or lactation
* Recently decompensated medical illness necessitating inpatient hospitalization (past 30 days)
* Transaminases (aspartate aminotransferase/alanine aminotransferase) greater than five times the upper limit of normal within 90 days of assessment phase
* Not well-controlled psychiatric symptoms at the time of physician assessment, including suicidal ideation or untreated psychosis; or recently decompensated psychiatric illness necessitating inpatient hospitalization (past 30 days).
* Use of a moderate to strong CYP3A4 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Becker, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Identify potentially eligible individuals that are prescribed an active opioid of 30-100mg. Patients are screened through medical records and referral from primary care providers in addition to a opt out letter and follow up phone call.
Period: Overall Study
Arm/Group | Buprenorphine/Naloxone | Opioid Dose Escalation
Started | 3 (3 patients were enrolled in the Buprenorphine arm of the study) | 4 (4 patients were enrolled in the opioid dose escalation arm of the study)
Completed | 1 (1 patient completed the Buprenorphine arm of the study. 2 patients withdrew) | 4 (4 patients completed the opioid dose escalation arm of the study)
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants were recruited and enrolled at VACT West Haven, CT. Participants are aged 18 and older and have 3 months or more of continuous opioid therapy for chronic pain. Participants are actively prescribed 30-100mg of morphine equivalent opioid dose based on pharmacy records. Primary Care Providers will assent for patient participation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine/Naloxone | Opioid Dose Escalation | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants] — We will measure a range of pre-treatment variables at baseline to ensure that participants meet eligibility criteria. Using validated instruments during treatment and at the end of treatment, we will examine the differential impact of BUP/NX versus opioid dose escalation including outcome assessments related to pain severity, pain interference and patient global assessment of change during treatment.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 1 | 1
    >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (4.6) | 69.8 (9.5) | 68.6 (7.4)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Numeric Rating Scale of Pain Severity
Description: Validated 11 pt scale 0-10, to evaluate a patient's current severity of pain. A rating of 0 indicates no pain while 10 indicates the worst pain imaginable. A score of 4 or above is considered a clinically significant pain level according to VHA treatment guidelines.
Time Frame: Baseline and 12 wks
Population: This group of subjects consisted of five males. One Buprenorphine subject aged-72 and four Opioid Dose Escalation subjects aged- 66,77,78,and 58.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine/Naloxone | Opioid Dose Escalation
Number analyzed (Participants) | 1 | 4
units on a scale | -2 (NA) — Not able to calculate a standard deviation. 1 subject completed this arm of the study. | 0.5 (1)

2. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The "Patient Global Impression of Change Scale" (PGIC) is one question capturing the individual's overall perception of efficacy of treatment in a clinical trial. It uses verbal outcome categories on a 7-point scale with "very much worse" and "very much better" as anchors and "no change" in the middle. The verbal categories were coded on a scale with -3 "very much worse",+3 "very much better", and 0 "same". To calculate the mean and standard deviation of each group (Bup/Opioid Increase) we took the sum of each participants final PGIC score and divided by the total number of participants.
Time Frame: 12 wks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine/Naloxone | Opioid Dose Escalation
Number analyzed (Participants) | 1 | 4
units on a scale | 1 (NA) — Not able to calculate a standard deviation. 1 subject completed this arm of the study. | 1 (1.15)

ADVERSE EVENTS:
Arm/Group | Buprenorphine/Naloxone | Opioid Dose Escalation
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

LIMITATIONS AND CAVEATS:
Aim 1 of the study was achieved: we found that despite moderate to high levels of pain interference, only a small proportion of eligible patients entered the trial. For this reason, the data & safety monitoring board recommended early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes